CLINICAL TRIAL: NCT03243669
Title: High Definition Endoscopy and Virtual Chromoendoscopy Versus Standard Resolution Endoscopy in Detection of Colon Polyps
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: S52580
Record Dates: First submitted 2017-07-22; First posted 2017-08-09 (Actual); Last update posted 2023-01-27 (Actual); Status verified 2017-08

CONDITIONS: Colonic Adenoma
Keywords: Colonoscopy; High-definition endoscopy; Virtual chromoendoscopy; Adenoma detection rate (ADR)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (11):
- Fujinon standard (Active Comparator)
  Interventions: Diagnostic Test: Standard
- Fujinon HD (Active Comparator): Fujinon high-definition
  Interventions: Diagnostic Test: High-definition
- Fujinon HD + VC (Active Comparator): Fujinon high-definition + virtual chromoendoscopy
  Interventions: Diagnostic Test: High-definition; Diagnostic Test: Virtual chromoendoscopy
- Olympus standard (Active Comparator)
  Interventions: Diagnostic Test: Standard
- Olympus HD (Active Comparator): Olympus high-definition
  Interventions: Diagnostic Test: High-definition
- Olympus VC (Active Comparator): Olympus virtual chromoendoscopy
  Interventions: Diagnostic Test: Virtual chromoendoscopy
- Olympus HD + VC (Active Comparator): Olympus high-definition + virtual chromoendoscopy
  Interventions: Diagnostic Test: High-definition; Diagnostic Test: Virtual chromoendoscopy
- Pentax standard (Active Comparator)
  Interventions: Diagnostic Test: Standard
- Pentax HD (Active Comparator): Pentax high-definition
  Interventions: Diagnostic Test: High-definition
- Pentax VC (Active Comparator): Pentax virtual chromoendoscopy
  Interventions: Diagnostic Test: Virtual chromoendoscopy
- Pentax HD + VC (Active Comparator): Pentax high-definition + virtual chromoendoscopy
  Interventions: Diagnostic Test: High-definition; Diagnostic Test: Virtual chromoendoscopy

INTERVENTIONS:
Diagnostic Test: High-definition — High-definition colonoscopy
  Arms: Fujinon HD; Fujinon HD + VC; Olympus HD; Olympus HD + VC; Pentax HD; Pentax HD + VC
Diagnostic Test: Virtual chromoendoscopy — Virtual chromoendoscopy
  Arms: Fujinon HD + VC; Olympus HD + VC; Olympus VC; Pentax HD + VC; Pentax VC
Diagnostic Test: Standard — Standard colonoscopy
  Arms: Fujinon standard; Olympus standard; Pentax standard

SUMMARY:
Over the last years a number of new endoscopic imaging modalities have been introduced (high-definition and virtual chromoendoscopy). Given the theoretical advantage of these new imaging techniques, the investigators aimed to investigate their use for the detection of polyps during colonoscopy.

ELIGIBILITY:
Inclusion Criteria:

* referred for colonoscopy
* signed informed consent

Exclusion Criteria:

* subtotal colectomy
* known colorectal tumor or polyp prior to colonoscopy
* genetic predisposition to colon cancer namely FAP, HNPCC, Hyperplastic polyposis syndrome, juvenile polyposis, Peutz-Jeghers syndrome
* inflammatory bowel disease
* primary sclerosering cholangitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2146 (Actual)
Dates: Start 2010-12-01 (Actual); Primary Completion 2014-06-30 (Actual); Study Completion 2014-12-31 (Actual)

PRIMARY OUTCOMES:
Adenoma detection rate (ADR) | 7-10 days
  Percentage of colonoscopies with detection of 1 or more adenomas. ADR is a well-established quality indicator in colonoscopy in the prevalence of adenomas detected (ADR) as recommended by American Society for Gastrointestinal Endoscopy (ASGE)/American College of Gastroenterology Task Force (ACGTF) and European Society of Gastrointestinal Endoscopy (ESGE). Guidelines stipulate to use ADR as main quality indicator in colonoscopy.

SECONDARY OUTCOMES:
Number of adenomas | 7-10 days
  Adenoma per colonoscopy rate (APCR)
Type of adenomas | 7-10 days
  Subtypes of adenomas: tubular adenomas, tubulovillous adenomas, sessile serrated adenomas and adenocarcinomas

CONTACTS AND LOCATIONS:
Overall Officials: Raf Bisschops, MD PhD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- University Hospitals Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rex DK, Schoenfeld PS, Cohen J, Pike IM, Adler DG, Fennerty MB, Lieb JG 2nd, Park WG, Rizk MK, Sawhney MS, Shaheen NJ, Wani S, Weinberg DS. Quality indicators for colonoscopy. Am J Gastroenterol. 2015 Jan;110(1):72-90. doi: 10.1038/ajg.2014.385. Epub 2014 Dec 2. No abstract available. PMID 25448873
- [Background] Kaminski MF, Thomas-Gibson S, Bugajski M, Bretthauer M, Rees CJ, Dekker E, Hoff G, Jover R, Suchanek S, Ferlitsch M, Anderson J, Roesch T, Hultcranz R, Racz I, Kuipers EJ, Garborg K, East JE, Rupinski M, Seip B, Bennett C, Senore C, Minozzi S, Bisschops R, Domagk D, Valori R, Spada C, Hassan C, Dinis-Ribeiro M, Rutter MD. Performance measures for lower gastrointestinal endoscopy: a European Society of Gastrointestinal Endoscopy (ESGE) Quality Improvement Initiative. Endoscopy. 2017 Apr;49(4):378-397. doi: 10.1055/s-0043-103411. Epub 2017 Mar 7. PMID 28268235